CLINICAL TRIAL: NCT02294630
Title: Aerosolized Survanta in Neonatal Respiratory Distress Syndrome: Phase I/II Study
Brief Title: Aerosolized Surfactant in Neonatal RDS
Acronym: AS-02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sood, Beena G., MD, MS (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1206011023; 1R01FD004793-01A1 (FDA); FD004793 (Other: FDA - OOPD)
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Surface-Active Agents; beractant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Schedule I (Active Comparator): Surfactant dose to be administered as aerosol - 100 mg phospholipid/kg. Surfactant Dilution 1:1
  Interventions: Drug: Surfactant
- Dose Schedule II (Active Comparator): Surfactant dose to be administered as aerosol - 100 mg phospholipid/kg. Surfactant Dilution 1:2
  Interventions: Drug: Surfactant
- Dose Schedule III (Active Comparator): Surfactant dose to be administered as aerosol - 200 mg phospholipid/kg. Surfactant Dilution 1:1
  Interventions: Drug: Surfactant
- Dose Schedule IV (Active Comparator): Surfactant dose to be administered as aerosol - 200 mg phospholipid/kg. Surfactant Dilution 1:2
  Interventions: Drug: Surfactant

INTERVENTIONS:
Drug: Surfactant — Two doses of surfactant to be administered as aerosol will be tested - 100 mg phospholipid/kg and 200 mg phospholipid/kg. Each dose will be tested at two dilutions and with two nebulizers. Each enrolled infant may receive a maximum of two aerosol treatments of a single dilution with a single nebulizer.
  Other Names: Survanta

SUMMARY:
Respiratory distress syndrome (RDS), caused by surfactant deficiency, is the leading cause of mortality and morbidity in preterm infants. Intratracheal instillation, the only approved means of surfactant delivery, requires endotracheal intubation and mechanical ventilation with their attendant risks. Interventions that decrease need for intubation and mechanical ventilation like noninvasive ventilation (NIV) including nasal continuous positive airway pressure, high flow nasal cannula or nasal intermittent mandatory ventilation are increasingly being used for initial respiratory support in preterm neonates with RDS to improve outcomes. Aerosolized surfactant delivered during NIV is an innovative and promising concept for the treatment of RDS - retaining the advantages of early surfactant with alveolar recruitment while obviating the risks of intubation and mechanical ventilation. The investigators overall hypothesis is that treatment of RDS with aerosolized surfactant in preterm infants undergoing NIV is safe and feasible and will result in short-term improvement in oxygenation and ventilation. The objective of this proposal is to perform a single-center unblinded Phase II randomized clinical trial of aerosolized surfactant for the treatment of RDS in preterm neonates undergoing NIV. Funding Source - FDA-OOPD.

ELIGIBILITY:
Inclusion Criteria:

1. Infants admitted to the NICU at Hutzel Women's Hospital (HWH)/Children's Hospital of Michigan (CHM)
2. Gestational age of 240/7-366/7 weeks
3. Postnatal age ≤ 24 hours
4. Clinical diagnosis of RDS based on (i) presence of at least two of the four classic symptoms (need of supplemental oxygen, tachypnea, intercostal retractions or grunting), and (ii) exclusion of other causes of respiratory failure and (iii) Clinician intent to administer surfactant if infant requires intubation
5. Respiratory support with NIV (CPAP or NIPPV or HFNC) with FiO2 ≥25% or PEEP ≥ 4 cmH20 or HFNC rate ≥ 2 LPM for ≤8 hours
6. Written informed consent from parent/guardian

Exclusion Criteria:

1. Previous receipt of surfactant
2. Infants with respiratory distress who are unstable and require immediate intubation
3. Active air leak syndrome (e.g. pneumothorax, pneumomediastinum)
4. Lethal congenital malformations; death anticipated within first 3 days of life; decision to withhold support
5. Serious abdominal, cardiac, airway or respiratory malformations including tracheal esophageal fistula, intestinal atresia, omphalocele, gastroschisis, pulmonary hypoplasia, or diaphragmatic hernia
6. Neuromuscular disorder resulting in respiratory compromise

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2014-12; Primary Completion 2019-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beena G. Sood, MD, MS, Principal Investigator — Wayne State University
Locations (1):
- Hutzel Women's Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Sood BG, Cortez J, Kolli M, Sharma A, Delaney-Black V, Chen X. Aerosolized surfactant in neonatal respiratory distress syndrome: Phase I study. Early Hum Dev. 2019 Jul;134:19-25. doi: 10.1016/j.earlhumdev.2019.05.005. Epub 2019 May 20. PMID 31121339
- [Result] Sood BG, Thomas R, Delaney-Black V, Xin Y, Sharma A, Chen X. Aerosolized Beractant in neonatal respiratory distress syndrome: A randomized fixed-dose parallel-arm phase II trial. Pulm Pharmacol Ther. 2021 Feb;66:101986. doi: 10.1016/j.pupt.2020.101986. Epub 2020 Dec 16. PMID 33338661

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 159 enrolled and randomized participants, 149 met eligibility criteria and proceeded with treatment.
Groups:
- Dose Schedule I; Dose Schedule III: Surfactant dose to be administered as aerosol - 100 mg phospholipid/kg.
  Surfactant: Two doses of surfactant to be administered as aerosol will be tested - 100 mg phospholipid/kg and 200 mg phospholipid/kg. Each dose will be tested at two dilutions and with two nebulizers. Each enrolled infant may receive a maximum of two aerosol treatments of a single dilution with a single nebulizer.
- Dose Schedule II; Dose Schedule IV: Surfactant dose to be administered as aerosol - 200 mg phospholipid/kg.
  Surfactant: Two doses of surfactant to be administered as aerosol will be tested - 100 mg phospholipid/kg and 200 mg phospholipid/kg. Each dose will be tested at two dilutions and with two nebulizers. Each enrolled infant may receive a maximum of two aerosol treatments of a single dilution with a single nebulizer.
Period: Overall Study
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Started | 37 | 38 | 35 | 39
Completed | 37 | 38 | 35 | 39
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV | Total
Number analyzed (Participants) | 37 | 38 | 35 | 39 | 149
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 31.4 (3.0) | 31.6 (3.3) | 31.0 (3.0) | 31.7 (3.2) | 31.4 (3.1)
Age, Customized [Count of Participants; unit: Participants]
  GA strata: GA strata I (24-28 weeks) | 7 | 7 | 8 | 7 | 29
  GA strata: GA strata II (29-32 weeks) | 16 | 15 | 14 | 15 | 60
  GA strata: GA strata III (33-36 weeks) | 14 | 16 | 13 | 17 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 20 | 14 | 78
  Male | 17 | 14 | 15 | 25 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 37 | 35 | 33 | 36 | 141
  Unknown or Not Reported | 0 | 1 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 38 | 35 | 39 | 149

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Feasibility
Description: Since surfactant reflux is typically considered to be one of the most likely adverse events associated with the intervention, it was planned to report the number of participants specifically with surfactant reflux for this Outcome Measure
Time Frame: During and within 6 hours after end of study drug administration, expected maximum of approximately 14 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants | 3 | 8 | 4 | 12

2. Primary Outcome: Patient Status as Evaluated by Dose Level
Description: Optimal dosing schedule was determined by preliminary evidence of efficacy (Need for intubation within 72 hours), lack of adverse effects, and overall infant comfort as assessed by bedside clinical caregivers.
Time Frame: During study drug administration, expected maximum of approximately 8 hours for adverse effects and infant comfort; need for intubation was assessed within 72 hours of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants
  Need for Intubation within 72 hours | 3 | 3 | 5 | 4
  Adverse events - surfactant reflux | 3 | 8 | 4 | 12
  Overall infant comfort during AS as assessed by bedside nurse (infant most comfortable) | 30 | 27 | 26 | 26

3. Primary Outcome: Short Term Efficacy as Assessed by Need for Intubation
Description: It will be suggested that infants be intubated and receive MV if they met 2 or more of 5 failure criteria: i). worsening clinical signs of respiratory distress (increasing tachypnea; expiratory grunting; intercostal, subcostal, and/or sternal recession); ii). apnea treated with positive pressure ventilation (PPV) by mask on 2 or more occasions in 1 hour; iii). FIO2 >0.5 to maintain pulse oxygen saturations 90%-95% for >30 minutes; iv). pH <7.2 on 2 arterial or capillary blood gases taken >30 minutes apart; and v). partial pressure of CO2 (PCO2) of >65 mm Hg on 2 CBG/ABGs taken 30 minutes apart.
Time Frame: Within 72 hours of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants | 3 | 3 | 5 | 4
Statistical Analysis 1: Comparison: Dose Schedule I vs Dose Schedule II; Test type: Other; p = 0.399, t-test, 2 sided

4. Secondary Outcome: Blood Gas Parameters - pH
Description: Blood gas pH
Time Frame: 60±30 minutes after end of study intervention
Measure: Mean (Standard Deviation); unit: pH units for pH, mmHg for pCO2
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 34 | 39
pH units for pH, mmHg for pCO2 | 7.35 (0.05) | 7.36 (0.07) | 7.36 (0.06) | 7.35 (0.05)

5. Secondary Outcome: Blood Gas Parameters - pCO2
Description: Blood gas pCO2.
Time Frame: 60±30 minutes after end of study intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
mmHg | 45 (8) | 45 (9) | 43 (6) | 45 (7)

6. Secondary Outcome: Pulse Oximetry
Description: Transcutaneous Pulse oximetry
Time Frame: 60±30 minutes after end of study intervention
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
percentage of oxygen saturation | 95.95 (3.34) | 96.95 (5.22) | 97.37 (3.16) | 97.47 (3.07)

7. Secondary Outcome: Vital Signs - Heart Rate
Description: Vital signs included heart rate, respiratory rate and systolic blood pressure
Time Frame: 60±30 minutes after end of study intervention
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
beats/minute | 134 (12) | 142 (14) | 138 (12) | 136 (12)

8. Secondary Outcome: Vital Signs - Respiratory Rate
Description: Vital signs included heart rate, respiratory rate and systolic blood pressure
Time Frame: 60±30 minutes after end of study intervention
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
breaths/minute | 47 (17) | 47 (15) | 46 (15) | 47 (15)

9. Secondary Outcome: Vital Signs - Systolic Blood Pressure
Description: Systolic blood pressure
Time Frame: 60±30 minutes after end of study intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
mmHg | 54 (9) | 51 (8) | 54 (10) | 53 (9)

10. Secondary Outcome: Number of Doses of Surfactant - Aerosolized & Intratracheal
Time Frame: Within 72 hours of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants
  One dose of aerosolized surfactant | 10 | 14 | 13 | 14
  Two doses of aerosolized surfactant | 27 | 24 | 22 | 25
  No. of doses of intratracheal surfactant - one | 0 | 2 | 2 | 0
  No. of doses of intratracheal surfactant - two | 2 | 0 | 1 | 1
  No. of doses of intratracheal surfactant - three | 0 | 0 | 1 | 2
  No. of doses of intratracheal surfactant - four | 0 | 1 | 0 | 0

11. Secondary Outcome: Pneumothorax, Pneumomediastinum or Other Air Leak
Time Frame: Within 72 hours of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants | 0 | 1 | 0 | 1

12. Secondary Outcome: Changes in Cerebral Oxygenation From Baseline as Evaluated at End of Study Intervention
Description: Changes in cerebral oxygenation from baseline as evaluated at end of study intervention
Time Frame: During and within 6 hours after end of study intervention, expected maximum of approximately 14 hours
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 35 | 36 | 33 | 38
percentage of oxygen saturation | 79 (8) | 80 (8) | 78 (11) | 79 (8)

13. Secondary Outcome: Changes in Surfactant Activity in Gastric Aspirates
Description: Concentration of major surfactant lipid (PC 16:0/16:0)
Time Frame: During study intervention, expected maximum of approximately 8 hours
Measure: Mean (Standard Deviation); unit: ng per mg of protein
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 22 | 24 | 22 | 23
ng per mg of protein | 10.9 (14.6) | 9.5 (9.2) | 8.8 (7.8) | 8.0 (8.0)

14. Secondary Outcome: Cumulative Duration of Non-invasive and Invasive Ventilation
Description: Cumulative duration of non-invasive and invasive ventilation at discharge
Time Frame: at discharge
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
number of days
  Duration of NIV (days) | 4.5 (8.1) | 7.0 (14.6) | 7.9 (14.2) | 6.1 (14.7)
  Duration of Invasive ventilation (days) | 1.3 (5.1) | 0.9 (4.0) | 1.6 (5.1) | 2.2 (7.4)

15. Secondary Outcome: Duration of Supplemental Oxygen, Intensive Care, Hospital Stay
Description: Duration of supplemental oxygen, and hospital stay
Time Frame: During initial hospital stay, expected <= 120 days
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
number of days
  Duration of supplemental oxygen (days) | 7.4 (18.5) | 9.0 (22.9) | 10.7 (25.2) | 8.9 (29.3)
  Length of hospital stay (days) | 29.9 (28) | 26.4 (24.3) | 32.1 (29.9) | 28.3 (30.8)

16. Secondary Outcome: Age at Start of Feeds, Feeding Progression, Age at Full Enteral Feeds
Description: Age at start of feeds, and age at full enteral feeds presented in days
Time Frame: During initial hospital stay, expected 1st 2 weeks of life
Measure: Mean (Standard Deviation); unit: age in days
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 36 | 34 | 39
age in days
  Age at start of feeds (days) | 1.3 (.7) | 1.6 (1.7) | 1.8 (1.7) | 1.5 (1.1)
  Age at full enteral feeds (days) | 11.2 (8.8) | 7.8 (7.3) | 11.8 (11.7) | 12.9 (12.9)

17. Secondary Outcome: Need for Blood Transfusions
Description: Number of infants requiring blood transfusions
Time Frame: During initial hospital stay, expected <= 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants | 10 | 6 | 8 | 7

18. Secondary Outcome: Growth Parameters
Description: Weight at discharge
Time Frame: At 7 days, 28 days, 36 weeks corrected GA and discharge
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
grams | 2153 (458) | 2222 (431) | 2235 (561) | 2281 (522)

19. Secondary Outcome: Morbidities Associated With Prematurity
Description: Grade III & IV IVH PDA requiring ligation ROP treated with Laser Surgical NEC BPD
Time Frame: During initial hospital stay, expected <= 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants
  Grade III & IV IVH | 0 | 1 | 0 | 1
  PDA requiring ligation | 0 | 1 | 0 | 0
  ROP treated with Laser | 0 | 1 | 0 | 1
  Surgical NEC | 0 | 0 | 2 | 2
  BPD | 4 | 4 | 5 | 2

20. Secondary Outcome: Survival to Hospital Discharge
Description: Survival to hospital discharge
Time Frame: During initial hospital stay, expected <= 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants | 37 | 38 | 35 | 39

21. Secondary Outcome: Survival to Discharge Without Severe Morbidity
Description: Survival to discharge without severe BPD, severe IVH, surgical NEC or ROP treated with Laser
Time Frame: During initial hospital stay, expected <= 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
Number analyzed (Participants) | 37 | 38 | 35 | 39
Participants | 37 | 35 | 33 | 35

ADVERSE EVENTS:
Time Frame: During and within 6 hours after the end of study drug administration, an expected maximum of approximately 14 hours
Arm/Group | Dose Schedule I | Dose Schedule II | Dose Schedule III | Dose Schedule IV
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38 | 0/35 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38 | 0/35 | 0/39
Other Adverse Events (participants affected / at risk) | 8/37 | 18/38 | 12/35 | 20/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Schedule I (N=37) | Dose Schedule II (N=38) | Dose Schedule III (N=35) | Dose Schedule IV (N=39)
Surfactant reflux from nose/mouth (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 4 | 12 — Surfactant reflux from nose/mouth
Desaturations (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 7 — Desaturations
Plugging of nasal prongs (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 — Plugging of nasal prongs
Increased secretions requiring suctioning (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 2 | 0 — Increased secretions requiring suctioning
Residual surfactant in nasal prongs (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 — Residual surfactant in nasal prongs
Dislodged prongs (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 — Dislodged prongs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT02294630/Prot_SAP_000.pdf